# Dynamics of Inflammation and its Blockade on Motivational Circuitry in Depression

Date: 11/26/2019

NCT03006393

IRB00087941

### You Are Being Asked to Be in a Research Study

Document Approved On: «ApproveDate»

Version Date: 11262019\_Mod20

### What Is a Research Study?

The main purpose of research studies is to gain knowledge. This knowledge may be used to help others. Research studies are not intended to benefit you directly, though some might.

#### **Do I Have to Do This?**

No. Being in this study is entirely your choice. If you decide to join this study, you can change your mind later on and withdraw from the research study.

Taking part in a study is separate from medical care. The decision to join or not join the research study will not affect your status as a patient.

#### What Is This Document?

This form is an informed consent document. It will describe the study risks, procedures, and any costs to you.

This form is also a HIPAA Authorization document. It will describe how your health information will be used and by whom.

Signing this form indicates you are willing to take part in the study and allow your health information to be used.

### What Should I Do Next?

- 1. Read this form, or have it read to you.
- 2. Make sure the study doctor or study staff explains the study to you.
- 3. Ask questions (e.g., time commitment, unfamiliar words, specific procedures, etc.)
- 4. If there will be medical treatment, know which parts are research and which are standard care.
- 5. Take time to consider this, and talk about it with your family and friends.

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


## Emory University Consent to be a Research Subject / HIPAA Authorization

Title: Infliximab

Study No.: «ID»

**Principal Investigator:** Michael Treadway, PhD

**Sponsor:** National Institute of Mental Health (NIMH)

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### What is the purpose of this study?

You are being asked to volunteer for a research study because you have been diagnosed with major depression or because you are participating as a healthy volunteer. The main purpose of this study is to examine the effects of a medicine called infliximab on measures related to depression symptoms. Infliximab is also known by its brand name Remicade. Infliximab, or Remicade, is given to people by an IV needle. It is currently used to treat two illnesses: rheumatoid arthritis and Crohn's disease. Infliximab is thought to help these conditions because it reduces inflammation in the body. Infliximab (Remicade) reduces inflammation by blocking a chemical in the body called tumor necrosis factor (TNF)-alpha. This chemical produces inflammation. Inflammatory chemicals in the body like TNF-alpha appear to be increased in some people with major depression. Researchers think that a drug like infliximab, which blocks TNF-alpha, may be helpful in treating depression. The Food and Drug Administration has not approved infliximab for treating depression. We plan to enroll up to 140 participants for this study.

Note: In some cases we will use a medicine similar to Infliximab in its place. This medicine, Inflectra, is an Infliximab biosimilar. This means that Inflectra is very similar to Infliximab but is not identical. While there may be some small differences between Inflectra and Infliximab, there are no clinically important differences in terms of safety and purity of the medicine. Inflectra is approved by the FDA for the same conditions as Infliximab. Please note each time you see Infliximab mentioned in this form, that Inflectra may be used instead.

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»


#### What will I be asked to do?

All procedures that you will be involved with in this study are experimental, except for the drawing of blood for routine laboratory tests to make sure you are not having a bad reaction to the study medicine.

Before you can participate in this study, you will need to come in for screening to see if you are able to enter the study. The investigator and/or the investigator's staff will ask you questions and run tests to determine if you are able to enter the study. These tests are described below. It is important that you answer all of the questions honestly and completely. If your condition or situation changes during the study, you must tell the investigator.

To be in this study, you must be off all antidepressant treatments for at least 8 weeks before the baseline visit. You cannot enroll in this study if you have had an antidepressant more recently than this period. If you are doing well on antidepressant medicine, you will not be able to be in this study. It would not be in your best interest to stop medicine that is helping you. If you have any questions or concerns about this, please speak with your physician or the study doctor.

You will not be able to enter the study if you are chronically taking a benzodiazepine at a dosage that is more than the equivalent of 2 milligrams a day of lorazepam.

If you plan to take any medicine or receive any medical treatment other than taking the study infusion given to you, please tell the study staff before starting the medicine or treatment. This includes medicines given to you or suggested by any other doctor. It also includes over-the-counter drugs. For example, cough treatments, cold treatments, pain medicines such as aspirin or ibuprofen, investigational drugs/procedures and sleeping medicines. If you plan to undergo elective surgery or a diagnostic procedure, you must tell the study staff before the procedure is performed.

You will be asked not to take the following medicines during the study:

- Aspirin
- Non-steroidal anti-inflammatory agents (such as ibuprofen or naproxen)
- COX-2 inhibitors (such as Celebrex or Bextra) during the study.

Use of these medicines may affect study findings. It is ok to use Tylenol during the study. However, please remember to tell the study staff if you've used this or any other medicines during the study. Please ask a study staff member if you are unsure if a medication you take falls in to one of the categories described above. You will receive a take-home instruction sheet that will remind you which medicines you should avoid while you are in this study. If you take one of these medications, whether on accident, out of necessity, or for any other reason, please contact the study team right away. The information sheet has contact information you can use to reach a member of the study staff. If you cannot reach the study team or need assistance after hours or on weekends/holidays, please call the Emory Clinic Operator at 404-778-5000 and ask them to page Bobbi Woolwine, LCSW at PIC# 15375. If you feel it is a medical emergency, please go to the nearest emergency room.

Although it is recommended that you do not drink alcoholic drinks during your participation in the study, you may drink alcohol on occasion (at most 1 glass of wine or equivalent per day). Use of illegal drugs during your participation in the study is not allowed. You will be drug-tested at each study visit for illegal drugs as part of this study.

If the study investigators (Dr. Treadway, Dr. Miller or their designees) decide that your depression has gotten worse at any time during the study, you may be asked to leave the study.

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


During this study you will interact with study investigators and doctors. You will also interact with research clinicians trained to administer psychiatric questionnaires and nurses trained to infuse drugs like infliximab. You will also interact with research coordinators who will help arrange your schedule during the study. A table of study events is provided below:

#### **Schedule of Visits**

| <u>Visit</u> | <u>Visit Overview</u> |
|---|---|
| Pre-Screening Visit | <ul> <li>Self-report questionnaires</li> <li>Blood work and/or finger stick</li> </ul> |
| Screening Visit(s) | <ul> <li>Clinical interview</li> <li>Self-report questionnaires</li> <li>Behavioral tasks</li> <li>Chest X-Ray</li> <li>EKG</li> <li>Laboratory testing</li> <li>Blood work</li> <li>Urine test</li> <li>Urine pregnancy test (if applicable)</li> <li>Urine drug test *Note that assessments completed during one Screening Visit will not be repeated at another. However, assessments will be repeated if deemed necessary under PI and/or study physician advisement. *Note that healthy controls will undergo all pre-screening and screening procedures as subjects, except that they will not receive a Chest X-Ray, EKG, or Quantiferon Gold TB Test</li> </ul> |
| Optional Scan Visit | <ul> <li>Behavioral tasks</li> <li>MRI Scan</li> <li>Blood work</li> <li>Urine drug test</li> <li>Urine pregnancy test (if applicable)</li> </ul> |
| Infusion Visit | <ul> <li>Clinical interview</li> <li>Self-report questionnaires</li> <li>Medical follow-up (F/U) assessment</li> <li>Laboratory testing</li> <li>Behavioral tasks</li> <li>Blood work</li> <li>Urine test</li> <li>Urine drug test</li> <li>MRI scan (if not performed previously)</li> <li>Infliximab or Placebo (salt water) Infusion</li> </ul> |

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


#### **Schedule of Visits (continued)**

| Optional 24 Hour Visit | <ul> <li>Clinical interview</li> <li>Self-report questionnaires</li> <li>Medical F/U assessment</li> <li>Blood work</li> <li>Vital signs</li> <li>Urine drug test</li> <li>Urine pregnancy test (if applicable)</li> </ul> |
|---|---|
| 3 Day Visit | <ul> <li>Clinical interview</li> <li>Self-report questionnaires</li> <li>Medical F/U assessment</li> <li>Behavioral tasks</li> <li>Blood work</li> <li>Vital signs</li> <li>Urine drug test</li> <li>Urine pregnancy test (if applicable)</li> </ul> |
| Optional 7 Day Visit | <ul> <li>Clinical interview</li> <li>Self-report questionnaires</li> <li>Medical F/U assessment</li> <li>Behavioral tasks</li> <li>Blood work</li> <li>Vital signs</li> <li>Urine drug test</li> <li>Urine pregnancy test (if applicable)</li> </ul> |
| 14 Day Visit | <ul> <li>Clinical interview</li> <li>Self-report questionnaires</li> <li>Medical F/U assessment</li> <li>Laboratory testing</li> <li>Behavioral tasks</li> <li>Blood work</li> <li>Vital signs</li> <li>Urine drug test</li> <li>Urine pregnancy test (if applicable)</li> <li>MRI scan</li> </ul> |

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


30 Day Phone Call

• Clinical interview

Abbreviations: EKG – electrocardiogram, CXR – chest x-ray, MRI scan – magnetic resonance imaging scan

If you agree to be in the study, this is what will happen.

To be in this study, you will have to complete up to three screening visits for the study staff to review and verify your eligibility. At the first screening visit, we will ask you to complete a short questionnaire. We will also draw some of your blood to measure a marker of inflammation called C-reactive protein. This could also be done using a finger stick.

Over all of the study visits, we will draw about 67 teaspoons of blood.

The following procedures will happen at additional screening visits, depending on your schedule and study staff availability. A study clinician or trained study staff member will ask you some questions about your mental health and psychiatric treatment history. A study doctor or nurse will review your medical history with you and will also conduct a physical examination. You will receive an electrocardiogram (EKG) and a chest x-ray to make sure you have no heart abnormalities. Also, some of your blood will be drawn to check for any abnormalities that would exclude you for study participation. This includes testing for the human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV). You will be excluded from the study and referred to your primary care physician should you test positive for any of these abnormalities. At the screening visits, you will also complete some questionnaires and behavioral assessments.

**Note**: If you have previously participated in another research study from our group, you may not have to complete some of the procedures in this study described under "Pre-Screening" and "Screening" if the results are still valid from the previous study. For your safety, however, some of these procedures may need to be re-done.

A marker of inflammation called C-reactive protein will also be measured in your blood. You will also have a tuberculosis blood test. This test requires a small blood draw. If this test is positive for tuberculosis you will not be able to enter the study. The study investigator will recommend that you contact your primary care doctor for a referral to a TB specialist. You will be excluded from the study if you have TB and need INH treatment. You will also receive a pregnancy blood test at your first screening visit if you are a female. At following visits, you will receive a urine pregnancy test. You will be excluded from the study if you are pregnant. We will ask you, regardless of if you are a man or a woman, to complete a form about the birth control you and your partner will use during the study period. The screening process will take in total about 7-8 hours spread out over two-three visits. It will occur at the Emory Clinic Building A and/or B, 1327 Clifton Rd, the Emory Department of Psychology, and/or the Atlanta Clinical Translational Science Institute (ACTSI) in the Emory University Hospital. You are strongly encouraged to ask the study investigator or a member of the study staff questions about the results of your lab tests and other diagnostic procedures.

If you qualify for the study and choose to enroll you will participate in 6-8 visits across about 2 weeks (depending on scheduling and other factors). All study visits will take place at one or more of the following places at Emory: Emory Clinic Building A and B, 1327 Clifton Road, the Emory Department of Psychology, and/or the ACTSI in the Emory University Hospital. At all visits a study clinician will ask you questions about symptoms of depression using a standardized interview. You will also fill out several self-report questionnaires. These will ask about depressive symptoms and about the quality of your life. We will analyze your blood to see whether a decrease in depression after

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


the infliximab infusion is linked to a decrease in inflammation chemicals. On the day of the infusion and the follow-up at 14 days, you will start your visit either at the Emory Department of Psychology or Emory Clinic Building A or Building B. On these days you may also go to the outpatient area in the ACTSI. The infusion may occur at either the ACTSI in the Emory University Hospital, or an infusion center in Emory Clinic Building A. For screening and all other follow-up visits, you will begin your study visit either at the Emory Department of Psychology or Emory Clinic Building A or B. On these days you may also go with the study coordinator to other places in the Emory Clinic or Emory University Hospital, like Cardiology, if certain tests and procedures are scheduled for that visit. The infusion study visit (including MRI scan) will take about 7-8 hours If you complete the MRI scan and infusion at separate visits, those visits will be about 2-3 hours and 5-6 hours respectively. The study visits at 24 hours (optional), 3 days, and 7 days (optional) after infusion will take about 3 hours. The study visit at 14 days after infusion will take about 5 hours. At each of these visits your blood will be drawn to do routine laboratory checks and also for research purposes.

**Please note:** You may be asked to complete a blood draw at each visit. The study investigators, including the study physicians, may decide it is in your best interest—and in the interest of safety—to repeat a test or collect a new test.

At screening and other visits, you will be asked to supply about 10 tablespoons of urine in a special cup. We may use the urine sample you provide to do a test to look for the presence of drugs of abuse, such as marijuana, cocaine or heroin. A positive test for any of these drugs at screening will prevent you from being in the study. We will also use the urine sample from this cup to test for the presence of a urinary tract infection (UTI). A positive urine test for drugs or a UTI at any visit may be a reason for withdrawing you from this study.

After the urine sample is collected, we may send the sample to a partner laboratory at Emory to conduct some further tests. If the sample collected at screening is not sufficient or a sample cannot be collected at that visit, we may ask you for another sample at a following visit. The researchers in this partner lab may take the cells from your urine to create something called induced pluripotent stem cells (iPSC). Using certain techniques, researchers can "reprogram" adult cells from urine and other sources to act like embryonic stem cells. These cells can then be directed to develop into specific types of cells in the body, like those found in the brain. For more information on how the cells from your urine sample may be used for this purpose, please see the section "How samples and/or data might be used".

If the urine or blood sample we collect is not sufficient for the further testing we may conduct or if we do not ask you to provide a urine or blood sample at your visit, we may ask you if you are willing to return to the lab to provide a sample.

Our study team will measure your vital signs, including pulse and blood pressure. These will be recorded lying down and/or standing at most visits. Your height, weight, and waist circumference (girth) will be measured during screening and your infusion visits. Further, head circumference and size as well as eye prescription strength may be recorded in order to prepare for the MRI scan.

Given constraints of time and study staff availability, we may complete the MRI scan portion of the infusion visit one day before the scheduled infusion. This will also depend, when possible, on your preference for scheduling the visits.

At or after your screening visit(s), a study staff member may ask you if you are interested in completing further assessments for the study through a mobile application. If you are interested, we may ask you to download the mobile app and complete brief questionnaires and/or behavioral tasks. We may ask you to complete assessments 1-5 times per day after your screening visit through up to 2 weeks after your final follow-up visit. Your compensation for this component of the study will depend on how many assessments you complete and your choices and performance in the behavioral tasks through the app.

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»

At the study visit on the day of the infusion, you will be randomly assigned (similar to a flip of a coin) to receive either infliximab or placebo (an inactive compound). As part of the study you will receive one infusion. The placebo will be salt water. You have a one in two chance of receiving infliximab and a one in two chance of receiving placebo. If you receive infliximab, your dose will be 5 milligrams for every kilogram of your body weight. The infusion will occur after your Screening visits and will take place at either an infusion center at Emory Clinic Building A or the ACTSI. You will sit in a special chair and a trained nurse will place an intravenous (iv) needle in a vein in your arm. Some of your blood will be drawn through the IV for routine labs and for research purposes before you receive the infusion, as described above.

Neither you nor the study investigator will know whether you receive infliximab or placebo. This is because all subjects will receive their infusions from identical looking bags that have been specially prepared for the study. However, if a medical emergency occurs, the information about whether you received infliximab or placebo is available to the study investigator. The IV bags with either infliximab or placebo will be prepared in a separate room. The bag will be connected to the IV in your arm. It will take about 2 hours for the infusion to be completed. You will be monitored for any type of bad reaction, such as an allergic response, during the infusion and for about 10-20 minutes afterwards. The nurse at the center you receive the infusion or one of the nurses or doctors on the study team may ask you to stay longer if they think it is best for your safety.

During the infusion visit, a study nurse or doctor will review your medical history with you and also complete follow-up assessment. For example, the nurse or doctor may ask you if there has been any change in the medications you take. A trained study staff member will complete a clinical interview with you and ask you about any bad reactions to a study procedure. Your height, weight, and vital signs will be recorded again at this visit. You will be asked to supply about 4 tablespoons of urine in a special cup. This will test for the presence of drugs of abuse, such as marijuana, cocaine or heroin. A positive test for any of these drugs at screening will prevent you from participating in the study. A positive test at any other visits may be a reason for withdrawing you from this study. Also, you will be asked to supply about 4 tablespoons of urine in the same or a different cup that will be used to test for the presence of a urinary tract infection. You will also complete some questionnaires and behavioral tasks on a computer if there is time.

Before you receive the infusion, a nurse or doctor from the study team or infusion center may ask you to take a medicine that could help prevent a bad reaction from the study drug. The medicine(s) you may be asked to take would be Tylenol, Benadryl, and/or Pepcid.

If you have a bad reaction to the study drug, the nurses at the site you receive the infusion are trained to help you. The nurse would follow a special protocol that includes steps for stopping the infusion, giving you some oxygen, and giving you some medicine (Benadryl, Pepcid, and/or adrenaline).

Please ask the study nurse or doctor if you have any questions or concerns about the medicines you may be asked to take before or after the infusion. Any medicine you would be asked to take would be to help prevent or make better any symptoms you were having from the infusion.

At the infusion and 14-day visits, we will also do an MRI scan. The scanning session may include several different types of scans: structural, diffusion tensor imaging, MR spectroscopy (MRS), and functional scans. For this part of the visit, a study staff member will escort you to or meet you at the Facility for Education and Research in Neuroscience (FERN) on the Emory main campus. The MRI scan will last for about 90 minutes. Before the MRI scan, we will ask you some questions to make sure it is safe for you to have an MRI.

**Note:** Based on scheduling and your preference, the first MRI scan may be completed the day before the infusion visit.

To be scanned, you will be asked to remove all jewelry and other metal-containing objects (including credit cards). You will enter a large room where a powerful magnet is located. You will be asked to lie down on a narrow table and then

 IRB Form 04152016 Version Date: 11262019 Mod20

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»


you will be put in a small tunnel about 6 feet long and 2 feet in diameter. You will then be asked to lie as still as possible during the scan. You will be wearing headphones and a small mirror will be positioned above your head so you will be able to see out the end of the scanner. During scanning, you will hear a loud banging noise as the MRI machine takes pictures of your brain. This is normal. You will be given earplugs to make you more comfortable. If you feel uncomfortable at any point, the MRI scanner has a microphone and you can ask us to stop the scanning procedure without penalty.

You will be getting a scan for research purposes only. The research does not require health professionals to read the scan. The researchers are not qualified to interpret the images for healthcare purposes. Do not rely on the scan for clinical or diagnostic purposes. However, if the researchers have a question about something they see on the scan they will tell you, and ask you if you want the scan sent to a qualified health professional for review and any further medical treatment. You or your insurance company may have to pay for the review and any such treatment.

During the scan, we may ask you to rate certain things by pressing buttons on a box. For example, we may ask you to rate how you are feeling at the moment. We may also ask you to do one or more computer tasks while in the MRI scanner.

You will be able to hear and speak to the research staff at all times during the scan. If you become uncomfortable or want to stop the scan for any reason, just tell us. We will stop the scanning process immediately.

Visits at 24 hours (Optional), 3 days, 7 days (Optional), and 14 days post-infusion will involve completing questionnaires asking about symptoms and side effects. A nurse practitioner or trained study staff member may also ask you questions about your symptoms and any changes you may have experienced during the study. A nurse practitioner may also complete a physical examination with you. Each of these visits will require about 2-3 hours of your time. At each of these visits some of your blood will be drawn to do routine laboratory checks and also for research purposes.

At your study visit on the day of screening, infusion and at 3, 7 (Optional), and 14 days post infusion, you will also be asked to complete a series of decision-making tasks. On the infusion day and 14-day visits, you may complete some of these tasks while in the MRI scanner. The tasks will require you to select different options using different buttons. Some tasks will require you to make your responses very rapidly.

Around one month after the infusion, you will receive a follow-up phone call from a study staff member. He or she will ask you questions to make sure you have not had a bad reaction to anything that happened in the study.

Participants recruited as healthy controls will undergo a shortened version of the study protocol consisting of pre-screening and screening visits, as well as a scan visit. Healthy controls will go through a pre-screen and screening process that will consist of psychiatric evaluations, research and safety labs, and baseline assessments (clinician-rated assessments, self-reports, behavioral tasks). The pre-screening and screening procedures will be identical to those a subject goes through, except that a healthy control will not receive a Chest X-Ray, EKG, or Quantiferon Gold TB Test. Healthy controls will undergo a scan visit as well. It is important to note, however, that healthy controls will not receive any drug or any infusion.

#### How will the study medicine be provided?

The study medicine that you will take will be dispensed by the pharmacy and delivered to the principal investigator or study team member. The principal investigator or health care providers on his/her research team will provide the medicine to you. If you have questions about the medicine, you should ask one of the study doctors or either of the study nurses. If you have an urgent question or concern related to the study medicine after normal business hours, please contact the Emory Clinic operator

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


#### Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may be still be used for this study. Urine samples will be safely disposed of immediately after each drug or pregnancy test is completed. Dr. Michael Treadway, the primary investigator, will own the research blood samples drawn in this study. Any study samples collected at ACTSI or the Emory Medical Lab (EML) will be managed by that facility.

#### What are the possible risks and discomforts?

This study is designed to test the effects of a medicine called infliximab on measures related to depression symptoms. The use of infliximab to treat major depression has not been approved by the Food and Drug Administration. There is no information regarding side effects or serious reactions to infliximab in medically healthy patients who receive infliximab. Some side effects and more serious reactions to infliximab have been reported in patients receiving the medication medicine for the treatment of rheumatoid arthritis or Crohn's disease.

The Food and Drug Administration (FDA) issued a Black Box Warning for this medicine because patients in treatment with this product are at increased risk of infections. This includes a worsening of symptoms that may lead to hospitalization or death. Please read the possible side effects in the table on the next page.

#### **Possible Side Effects of Infliximab**

#### Other Important Risk Information to Consider

• Most of the possible rare side effects described in the table occurred in patients who were taking other

| Rare Side Effects (less than 1% of patients) | Occasional Side effects (1-10% of patients) | Frequent (10-50% of patients) |
|---|---|---|
| Severe immediate allergic reaction | Shortness of breath | Mild allergic reaction |
| Delayed allergic response to medicine | Itchy skin | Stomach pain |
| Serious bacterial infection | Chest pain | Nausea |
| Tuberculosis | An abscess | Diarrhea |
| Fungal infection | Insomnia | Heartburn |
| Death | Depression | Upper respiratory tract infection |
| | Oral thrush | Sore throat |
| | | Sinusitis (sinus infection) |
| | | Coughing |
| | | Runny nose |
| | | Rash |
| | | Fatigue |
| | | Fever |
| | | Headache |
| | | Joint pain |
| | | Back pain |
| | | Urinary tract infection |
| | | Hypertension |

medicines that suppress the immune system while they were taking infliximab. If you choose to enter this study

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»

you will be tested for tuberculosis using the Quantiferon Gold blood test. If this test is positive you will not be able to participate in the study.

- At screening you will be asked if you have any symptoms of infection or if you have a history of any chronic or serious infections. If you do, you will be excluded from the study.
- An increased risk of infection has been noted in patients taking drugs like infliximab who are also taking a drug called anakinra. If your doctor has prescribed anakinra for you, you will not be eligible for this study.

#### Possible Allergic/Delayed Reactions to Infliximab

| Symptoms of severe immediate allergic reaction | Symptoms of serious delayed reaction |
|---|---|
| Hives (red, raised, itchy patches of | Fever |
| skin) | |
| Difficulty breathing | Rash |
| Chest pain | Headache |
| High or low blood pressure | Muscle or joint pain |

Symptoms of severe immediate allergic reaction to infliximab can include hives (red, raised, itchy patches of skin), difficulty breathing, chest pain and high or low blood pressure. Symptoms of serious delayed reaction may include fever, rash, headache, and muscle or joint pain. If allergic symptoms occur during or immediately after the infusion you will be evaluated by a study physician who is expert at treating these symptoms. There is a standard procedure in place for treating allergic reactions at either of the locations you might receive the infusion. If you develop symptoms of a delayed reaction at home, or if you develop any of the negative health events listed above, you should contact the study clinician immediately. To do this, call the Emory Clinic operator (available 24 hours a day) at

. The study coordinator will give you an emergency information contact card to keep


in your wallet.

#### Congestive heart disease

- Infliximab has been reported to worsen a condition called congestive heart disease and to lead to increased deaths in patients with this condition. You will be asked about any history of heart disease.
- In addition, you will receive an electrocardiogram (EKG) at the Emory Clinic or ACTSI. This test checks if your heart is working normally.
- To be enrolled in this study, you will need to have a normal EKG and no history of heart disease.
- No known risks are connected to the EKG screening test. However, it is possible the gel or tape, used in the procedure, may cause skin irritation at the site of the electrode(s).

#### Decrease in white and red blood cells

- Infliximab has been rarely connected to a decrease in white and red blood cells, as well as platelets.
- There have been reports of death from these blood cell abnormalities in patients taking infliximab. However, it has not been proven that infliximab directly caused these abnormalities.
- You will have your blood cells examined before and after the infusion during the study. This test will occur at
  each assessment visit. If your red or white blood cells or platelets are abnormal before the infusion you will be
  excluded from the study.

#### Central nervous system conditions

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»


- In rare cases, Infliximab has been connected to a variety of central nervous system conditions. These include inflammation of the nerves of the eye, seizures or a condition like multiple sclerosis.
- The study investigator will ask you about any history of central nervous system disorders, such as multiple sclerosis or seizures. If you have a history of a central nervous system illness such as multiple sclerosis, Guillain-Barre syndrome or seizures, or have tingling or numbness in any part of your body, you will be excluded from study participation.

#### Allergic reaction to handling rodents and/or taking medicines made from mouse chemicals

- You will be asked if you have ever had an allergic reaction from being around, or handling rodents. If you have had such an allergic reaction you will not be able to be in this study.
- You will also be asked if you have ever had an allergic reaction to medicines made from mouse chemicals. These
  medicines include basiliximab (Simulect), daclizumab (Zenapax), gemtuzumab ozogamicin (Mylotarg), rituximab
  (Rituxan) and trastuzumab (Herceptin). These medicines are used for cancer and to stop transplanted organs
  from being rejected from the body. If you have ever had an allergic reaction to any of these medicines you will
  not be able to be in this study.

#### Autoimmune conditions

- Infliximab may increase the risk of developing an autoimmune condition like systemic lupus erythematosis or multiple sclerosis. But, this has not been proven.
- At screening you will be asked whether you have a history of any autoimmune related disorders, including lupus
  and multiple sclerosis. This also includes other conditions such as Crohn's disease, ulcerative colitis, rheumatoid
  arthritis, ankylosing spondilitis, scleroderma, thyroid or parathyroid disease or sarcoid.
- If you have a history of any autoimmune condition you will not be eligible for this study.

#### Live virus vaccines

- It is not known whether receiving infliximab would increase the risks involved in receiving a modified live virus
  vaccine. For this reason you will be asked about whether you have received a vaccine within four weeks of study
  entry.
- You will also be asked if you plan to receive a vaccine during the study or for a month afterwards. It is very important that you not receive any modified live virus vaccines for a month before the study, during the study and for at least one month after you have finished the study.
- You will not be able to be in this study if you have or will receive a vaccine during this time. Examples of common modified live virus vaccines include vaccines for smallpox (vaccinia), measles, mumps, rubella (MMR), varicella (chicken pox and shingles), yellow fever and the oral vaccines for: influnza (flu), typhoid, and polio vaccines. The injectable forms of influenza (flu), typhoid, and polio are killed (inactive) vaccines.

#### Cancer

- People who have been treated with Infliximab for rheumatoid arthritis or Crohn's disease for a long time tend to be more prone to a type of blood cancer called lymphoma.
- There have been some patients that while taking infliximab developed other types of cancer. But, the number of people taking infliximab that developed cancer does not seem to be much different from what you would expect to see in people who are not taking infliximab.
- It is not known whether brief treatment with infliximab is a risk for cancer in medically healthy subjects, such as in this study.
- If you have ever had any type of cancer in the past, including skin cancer, you will not be able to be in this study.

In addition to risks related to taking infliximab there are other risks linked to participating in this study.

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»


#### Other Risks

#### Drawing Blood and Finger Stick

- The risks of inserting and drawing blood from a finger stick, venous catheter or a syringe are minimal. The risks include swelling, tenderness, discomfort, bruising, infection, bleeding and fainting.
- To minimize these risks, the procedure will be done in a sterile manner by trained research or clinical staff while you are comfortably seated.
- Venous catheter placement and blood withdrawal will be done by nurses or trained phlebotomists with extensive experience with blood drawing.
- The amount of blood that we will draw over the course of the study is in compliance with the American Red Cross safety guidelines.

#### Psychiatric/Psychological Assessments

- The assessment of psychiatric and psychological issues may be connected to disturbing memories or feelings.
- To minimize this, you will be given ample opportunity during the assessment to discuss any disturbing memories or feelings you may experience.
- Research staff will be careful to avoid causing undue psychological distress during any part of the psychiatric assessment.

#### Computer Tasks/Cognitive Testing

- No known risks are linked to the computerized cognitive testing or computer tasks you will do.
- Some of the computerized tasks may be boring, but otherwise pose no risk.

#### Mobile App

You may be distracted in your daily life by phone notifications and/or email notifications to complete
assessments.

#### MRI

- The MRI machine is as loud as riding in a loud train you will be given earplugs and headphones to lessen the noise.
- You may experience some muscle discomfort while lying in the scanner.
- You may also become too hot or too cold, in which case you may ask for an adjustment of room temperature or a blanket.
- Some people become nervous or claustrophobic (anxious or afraid of closed spaces) in the scanner. If
  this happens to you, you may ask to be withdrawn immediately. You may also experience a sense of
  dizziness in the magnet. This is due to the strong magnetic field, and if it disturbs you, you may ask to be
  withdrawn.
- The magnetic field will affect any metallic object. You should not participate if you have any type of metallic implant in your body, including pacemakers, aneurysm clips, shrapnel, metal fragments, orthopedic pins, screws, or plates, non-MR safe IUD's (if you are unsure, you should discuss with study staff and/or your doctor), or piercings that you cannot remove. If you have any of these items in your body, there is a risk that the magnetic field could cause them to move or heat up. It is important that you inform the study staff if you have any implants.
- This type of brain scan is not designed to detect problems of the brain. You will be getting a scan for research purposes only. The research does not require health professionals to read the scan. The

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


researchers are not qualified to interpret the images for healthcare purposes. Do not rely on the scan for clinical or diagnostic purposes. However, if the researchers have a question about something they see on the scan they will tell you, and ask you if you want the scan sent to a qualified health professional for review and any further medical treatment. You or your insurance company may have to pay for the review and any such treatment.

#### Treatment for Depression

- Participation in this study will delay the delivery of active treatment for your depression.
- The risks connected to the delay of treatment for depression include continued symptoms of depression with the accompanying distress and difficulty in functioning, the possibility of worsening of the depressive symptoms, including the risk of suicidality.

The risk of suicide is always possible with depression. Please call the Emory Clinic operator at (404) 778-5000 and ask for Bobbi Woolwine, LCSW to be paged at #15375, immediately if you experience thoughts of suicide. If you feel that you are at risk of harming yourself, please go to the nearest emergency room.

#### Risks with Pregnancy

- The study medicine (infliximab or placebo) may involve currently unforeseeable risks to pregnant women, the embryo or fetus, or to children of nursing women.
- If you are a woman who is pregnant, breast feeding, or planning to become pregnant within the period of the study, you must not participate in the study. Also, all women of childbearing potential are required to undergo pregnancy testing before entering the study and at each study visit. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.
- All women of child bearing potential must use a medically acceptable contraceptive throughout the study. This
  includes oral (birth control pills), double-barrier method, injectable or implantable, or mechanical contraception.
  It also includes women whose sexual partners have had a vasectomy or have received or are using mechanical
  contraceptive devices. Condoms should be used in addition to other contraceptive methods to provide
  protection against sexually transmitted diseases and to provide added protection against pregnancy.
- All women of child bearing potential will be asked to abstain from sexual activity for 14 days prior to the study infusion visit.
- If you miss a period or think you might be pregnant during the study, you must tell the investigator immediately so that you can be withdrawn from the study.
- For women of childbearing potential, if you (a) plan to become pregnant, (b) become pregnant, (c) think you may have become pregnant, or (d) plan to discontinue contraception, you must tell the study investigator immediately.

**If you are a woman**: to protect against possible side effects of the study drug, women who are pregnant or nursing a child may not take part in this study. If you become pregnant, there may be risks to you, the embryo, or fetus.

**If you are a man:** the effect of the study drug on sperm is not known. You and the study doctor should agree on a method of birth control to use throughout the study. Men who are participating in this research study need to understand the possible danger of taking a drug that's effects on a fetus are unknown.

#### Study Drug

The study drug taken in this study may also have unknown risks.

Emory University IRB
IRB use only

Document Approved On: «ApproveDate»


#### **New Information**

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

#### Will I benefit directly from the study?

This is not a treatment study. Taking part in this research study may not benefit you personally, but researchers may learn new things about that treatment of depression that will help others. You will receive a single dose of the study drug as a part of this study. The study medicine may have no beneficial effect for you. Your depression may continue or worsen. You may benefit from this experimental research if the study medicine or placebo reduces your depressive symptoms. However, it is unlikely that you will benefit long-term from a single dose of the study drug, Infliximab. If you do benefit from a single dose of the study drug, it is unlikely that you will be able to continue to receive the drug outside of this study. Results from this study may also provide new understandings of the chemicals that are believed to be involved in major depression.

#### Will I be compensated for my time and effort?

To compensate for time required for participation, inconvenience and travel expenses, you will receive \$100, \$60, and \$200 for the outpatient study visits at 24 hours (Optional), 3 days, and 7 days (Optional) after your infusion respectively. You will receive \$100 for the pre-screening visit (which may be done prior to consent through the Behavioral Immunology Program), and \$100 for screening visit procedures. You will receive \$410 for the infusion visit, and \$310 for the study visit at 14 days (because you will receive an MRI scan at this visit). During the visits where you receive an MRI scan (on the day of infusion and at 14 days after infusion), you will have the opportunity to earn an additional \$150 per visit based on your choices and performance in a series of computer tasks. You may have the option of completing the MRI scan portion of the infusion visit one day before infusion. At visits on days 3 and 7 after infusion, you will have the opportunity to earn an additional \$50 per visit based on your task choices and performance. As a result, you will be compensated \$880 for this study but could earn up to \$1,580 total across all study visits. You will also receive a physical examination, EKG and laboratory evaluations free of charge as a result of participating in this study.

If you participate in the daily assessment part of this study, and complete all assigned days of assessment with the mobile app, you will receive an additional \$2-10 dollars for each day of mobile assessments you complete. The exact compensation you receive will be based on your choices and performance in the task(s) on the mobile app. If you complete 3 days of assessments, you could receive between \$6 and \$30. If you complete 7 days of assessments, you could receive between \$14 and \$70, and so on. You may earn up to \$150 for completing the mobile assessments. This would make your maximum amount of compensation across all visits \$1,730.

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»


| Visit | Total Amou | nt Earned |
|---|---|---|
| PRE-SCREENING (May be completed and compensated through Behavioral Immunology Screening Clinic) | \$100 | |
| Visit Total | | \$100 |
| SCREENING VISIT(S) | | |
| Visit A | \$50 | |
| Visit B | \$50 | |
| Visit Total | | \$100 |
| INFUSION VISIT(S) | | |
| fMRI (May be completed one day before infusion day) | \$250 | |
| Infusion | \$100 | |
| Scheduled Assessment | \$60 | |
| Visit Total | | \$410 |
| 24-HOUR VISIT (OPTIONAL) | | |
| Scheduled Assessments | \$100 | |
| Visit Total | | \$100 |
| 3-DAY VISIT | | |
| Scheduled Assessments | \$60 | |
| Visit Total | | \$60 |
| 7-DAY VISIT (OPTIONAL) | | |
| Scheduled Assessments | \$200 | |
| Visit Total | | \$200 |
| 14-DAY VISIT | | |
| fMRI | \$250 | |
| Scheduled Assessments | \$60 | 4 |
| Visit Total | | \$310 |
| TASK PERFORMANCE | 11.1.6450 | |
| Infusion Visit | Up to \$150 | |
| 3-Day Visit | Up to \$50 | |
| 7-Day Visit (OPTIONAL) | Up to \$50 | |
| 14-Day Visit Assessment Total | Up to \$150 | Up to \$400 |
| MOBILE APP (Optional) | | 3P to 3400 |
| Pre-Infusion Assessments (2 Days) | \$4-20 | |
| Post-Infusion Assessments (8 Days) | \$16-80 | |
| 80% Completion Bonus (8 of 10 Days) | \$50 | |
| Assessment Total | | Up to \$150 |
| Minimum Over Course of Study | \$880 | |
| Maximum Over Course of Study | \$1,830 | |

You may be paid by check or prepaid card. You will be asked to fill out a tax form, including your Social Security or Taxpayer Identification Number. If you elect payment via check, the check will be mailed to your house, which may be seen by others in your household. Depending on processing time, the compensation check may take up to about 4-6 weeks to arrive and will not be paid until after completion of the study. All payment for performance on tasks will be issued after completion of the study (regardless of payment method). The payment card is a prepaid debit card. It can be used exactly like a Mastercard. We load money onto your card electronically every time you need to be paid. The card scheme is run by Greenphire, an independent company specializing in payments for research studies and clinical trials. To issue your card, we need to give Greenphire some of your personal information. Banks and other financial institutions can access this information if they need to verify your identity when you use your card. Emory University is required by law to report any payments we make to the IRS. To do this, Emory University Department of Finance needs to keep your Social Security Number on file. We are asking you to allow us to communicate your name, address, date of birth,

Study No.: «ID» Emory University IRB
IRB use only

Document Approved On: «ApproveDate»


research study name and Social Security Number to Greenphire and Emory University Department of Finance. If you want to receive e-mail or text alerts when payments are made to you, we will ask you to provide your e-mail or phone number as well. All of this information will be stored on computers owned by Greenphire. Greenphire will not have access to any other information collected during this study. Full instructions about using your card are included when/if we issue it. Please ask if you have any questions or concerns about the card scheme or the use of your personal information.

#### What are my other options if I want treatment now?

Participation in this study does not include treatment. If you decide not to enter this study, there is care available to you outside of this research study.

Some medicines as well as other talking or behavioral therapies, which may be evaluated to treat your condition include, but are not limited to:

- Antidepressants (such as Paxil or Zoloft),
- Tricyclic antidepressants (including clomipramine),
- Monoamine Oxidase Inhibitors (such as phenelzine),
- Electroconvulsive shock therapy (ECT)
- Talking therapy (formal psychotherapy, and/or cognitive-behavioral therapy)

Participation in this study is not a substitute for your usual medical care by your regular doctor or specialist. At your request, we will give you copies of the results to review with your regular doctor or specialist.

The study investigator will discuss potential benefits and side effects of these treatments with you. You may choose to be treated with one or more of these treatments rather than participate in the study. Their effectiveness and side effects can vary according to their suitability for an individual patient. Some side effects include but are not limited to headache, sleepiness, diarrhea, insomnia, and sexual dysfunction. You do not have to participate in this research study to be treated for your condition.

Taking part in this study, however, may make you unable to participate in some other research studies, if they exclude people who have taken certain treatments. You should discuss this with the researchers if you have concerns. You may wish to research other study options at websites like clinicaltrials.gov and ResearchMatch.org.

#### How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

There is a Certificate of Confidentiality from the National Institutes of Health for this Study. The Certificate of Confidentiality helps us to keep others from learning that you participated in this study. Emory will rely on the Certificate of Confidentiality to refuse to give out study information that identifies you. For example, if Emory received a subpoena for study records, it would not give out information that identifies you.

The Certificate of Confidentiality does not stop you or someone else, like a member of your family, from giving out information about your participation in this study. For example, if you let your insurance company know that you are in this study, and you agree to give the insurance company research information, then the investigator cannot use the Certificate to withhold this information. This means you and your family also need to protect your own privacy.

The Certificate does not stop Emory from making the following disclosures about you:

**Emory University IRB** IRB use only

Study No.: «ID» Document Approved On: «ApproveDate»

- Giving state public health officials information about certain infectious diseases,
- Giving law officials information about abuse of a child, elderly person or disabled person.
- Giving out information to prevent harm to you or others.
- Giving the study sponsor or funders information about the study, including information for an audit or evaluation.

#### Storage and release of samples, genomic data, and health information

Portions of your samples, genomic data, and health information will be stored and shared with other researchers. The samples and information will be available for any research question, such as research to understand what causes certain diseases (for example heart disease, cancer, or psychiatric disorders), development of new scientific methods, or the study of where different groups of people may have come from.

#### How samples and/or data might be used:

We will use your samples and data only for research. We will not sell them. However, the results of this research might someday lead to the development of products (such as a commercial cell line, a medical or genetic test, a drug, or other commercial product) that could be sold by a company. You will not receive money from the sale of any such product. For more information on how your data may be shared with other researchers, please see the section called "National Institute of Mental Health Data Archive".

For this study, your samples and data will be used for purposes like making sure you are eligible to complete certain parts of the study like the MRI scans.

Your urine samples may be used to create a living tissue sample (called a "cell line") that can be grown in the laboratory. This allows researchers to have an unlimited supply of your cells in the future without asking for more samples from you.

We may use the cells taken from your urine to create a type of cell known as a pluripotent cell. This type of cell can be used to create different types of tissue, including cells found in the brain called neurons. Your cells might be used in research involving genetic alteration of the cells.

Your cells may be mixed with other human cells, mixed with animal cells, or grown in lab animals like mice.

What you should know about the cell lines that will be derived in the course of this study:

- The cell lines created will be similar or identical to you genetically.
- The cell lines may be kept indefinitely.
- There is the possibility that your cells or the created cell lines might be used in research that will involve genetic manipulation of the cells or the mixing of human and non-human cells in the animal models.
- The cell lines may be shared with researchers both inside and outside of Emory University, including commercial partners.
- The cell lines may be used to develop treatments for a variety of diseases and conditions.

#### National Institute of Mental Health Data Archive

Data from this study may be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share deidentified information with each other. A data repository is a large database where information from many studies is stored and managed. Deidentified information means that all personal information about research participants such as name, address, and phone number is removed and replaced with a code number. With an easier way to share, researchers hope to learn new and important things about mental illnesses more quickly than before.


Study No.: «ID» Emory University IRB
IRB use only

Document Approved On: «ApproveDate»


During and after the study, the researchers will send deidentified information about your health and behavior and in some cases, your genetic information, to NDA. Other researchers nationwide can then file an application with the NIMH to obtain access to your deidentified study data for research purposes. Experts at the NIMH who know how to protect health and science information will look at every request carefully to minimize risks to your privacy.

You may not benefit directly from allowing your information to be shared with NDA. The information provided to NDA may help researchers around the world treat future children and adults with mental illnesses so that they have better outcomes. NIMH will also report to Congress and on its web site about the different studies that researchers are conducting using NDA data. However, you will not be contacted directly about the data you contributed to NDA.

You may decide now or later that you do not want to share your information using NDA. If so, contact the researchers who conducted this study, and they will tell NDA, which can stop sharing the research information. However, NDA cannot take back information that was shared before you changed your mind. If you would like more information about NDA, this is available on-line at http://data-archive.nimh.gov.

#### How is my Genetic Information Protected? What are the Risks?

The Genetic Information Nondiscrimination Act (GINA) is a federal law that generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that GINA does <u>not</u> protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance, and does not apply to employers with less than 15 employees.

In addition to GINA, the State of Georgia has laws that prohibit insurers from using genetic testing information for any non-treatment purpose. However, like GINA, this state law protection has exclusions: life insurance policies, disability income policies, accidental death or dismemberment policies, medicare supplement policies, long-term care insurance policies, credit insurance policies, specified disease policies, hospital indemnity policies, blanket accident and sickness policies, franchise policies issued on an insurance policy written as a part of workers' compensation equivalent coverage, or other similar limited accident and sickness policies.

#### **Privilege**

In the State of Georgia, your genetic information has special legal protections called "privilege," which means that the information cannot be used as evidence in a court. By signing this form and allowing us to use and disclose your genetic information for the purposes described in this consent, you waive any privilege with regard to that genetic information, meaning that the information loses this legal protection.

#### What will happen to samples and/or data following a change in participation status:

If you decide to withdraw from the study, become ineligible to continue in the study, or have some other change in status that might affect your willingness to participate we might continue to use your stored samples and/or genomic data.

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»


#### What will happen to samples and/or data if the repository closes:

Your samples and/or genomic data will be transferred or destroyed if the repository closes.

#### **Medical Record**

We will take reasonable steps to keep copies of this form out of Emory Healthcare's medical records system. If we aren't successful in keeping these forms out, despite our efforts, we will take steps to remove them. If they cannot be removed, we will take steps to limit access to them.

Emory Healthcare may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your Emory Healthcare medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure.

The results of some study tests and procedures will be used only for research purposes and will *not* be placed in your medical record. For this study, those items include: the urine drug and urine and blood pregnancy tests, the research blood work, and the MRI scans.

Tests and procedures done at non-Emory places may not become part of your Emory medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.

#### In Case of Injury

If you get ill or injured from being in the study, Emory will help you get medical treatment. Emory and the sponsor have not, however, set aside any money to pay you or to pay for this medical treatment. The only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory or sponsor employee. "Negligence" is the failure to follow a standard duty of care.

If you become ill or injured from being in this study, your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurer does not pay, then you will have to pay these costs.

If you believe you have become ill or injured from this research, you should contact Dr. Michael Treadway at telephone number . You should also let any health care provider who treats you know that you are in a research study.

#### **Costs**

There will be no costs to you for participating in this study, other than basic expenses like transportation. You will not be charged for any of the research activities.

#### Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, if you leave the study before the final planned study visit, the researchers may ask you to have some of the final follow-up steps done.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

#### **Authorization to Use and Disclose Protected Health Information**

Emory University IRB IRB use only

Document Approved On: «ApproveDate»

The privacy of your health information is important to us. We call your health information that identifies you, your "protected health information" or "PHI." To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act and regulations (HIPAA). We refer to all of these laws as the "Privacy Rules." Here we let you know how we will use and disclose your PHI for the study.

#### PHI that Will be Used/Disclosed:

The PHI that we will use or share for the main research study includes:

- Medical information about you including your medical history and present/past medicines.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.
- Biological samples.
- Genetic information.
- Clinical records.

#### Purposes for Which Your PHI Will be Used/Disclosed:

We will use and share your PHI for the conduct and oversight of the research study. We will use and share your PHI to provide you with study related treatment and for payment for such treatment. We will also use and share your PHI to conduct normal business operations. We may share your PHI with other people and places that help us conduct or carry out the study, such as laboratories, data management centers, data monitors, contract research organizations, Institutional Review Boards (IRBs) and other study sites. If you leave the study, we may use your PHI to determine your health, vital status or contact information.

#### Use and Disclosure of Your Information That is Required by Law:

We will use and disclose your PHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults.

#### Authorization to Use PHI is Required to Participate:

By signing this form, you give us permission to use and share your PHI as described in this document. You do not have to sign this form to authorize the use and disclosure of your PHI. If you do not sign this form, then you may not participate in the research study or receive research-related treatment. You may still receive non-research related treatment.

 IRB Form 04152016 Version Date: 11262019\_Mod20

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


#### People Who will Use/Disclose Your PHI:

The following people and groups will use and disclose your PHI in connection with the research study:

| Person/Entity | <u>Purpose</u> |
|---|---|
| | To conduct the study entitled, "Dynamics of Inflammation and its Blockade on Motivational Circuitry in Depression", the purpose of which is to establish the validity of an inflammation-dependent path towards the development of motivational anhedonia. |
| _ | To monitor safety, efficacy and compliance with applicable laws and regulations. |
| University personnel, committees and departments charged with oversight of research, including the Institutional Review Board (IRB). | To monitor safety and compliance with applicable laws, regulations and University policies and procedures, and to run normal business operations. |
| Statisticians hired by the study sponsor. | To perform data analysis. |
| Emory University laboratories hired by the researchers | To analyze specimens. |

**Other:** Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your PHI may be shared with that new institution and their oversight offices. PHI will be shared securely and under a legal agreement to ensure it continues to be used under the terms of this consent and HIPAA authorization.

#### **Expiration of Your Authorization**

The Researchers will continue to use your PHI until the time at which the study is closed and the period for which any records relating to the study must be retained. After this, your Authorization to use your PHI will end and all identifiers will be removed from your information making it impossible to link you to the study.

#### Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them.

#### Emory University IRB IRB use only

Document Approved On: «ApproveDate»

To maintain the integrity of this research study, you generally will not have access to your PHI related to this research until the study is complete. When the study ends, and at your request, you generally will have access to your PHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you.

If it is necessary for your health care, your health information will be provided to your doctor. In general, we will not give you any individual results from the study of the samples you give us. If we find something of urgent medical importance to you, we will inform you, although we expect that this will be a very rare occurrence.

We may remove identifying information from your PHI. Once we do this, the remaining information will not be subject to the Privacy Rules. Information without identifiers may be used or disclosed with other people or organizations for purposes besides this study.

#### Other Items You Should Know

Dr. Treadway is a co-inventor of the EEfRT task software, which is used in this study. Emory University and Vanderbilt University licensed this software to BlackThorn Therapeutics. Under the IP Policies of both universities, Dr. Treadway receives licensing fees and royalties from BlackThorn Therapeutics. Additionally, Dr. Treadway has a paid consulting relationship with BlackThorn. The terms of this arrangement have been reviewed and approved by Emory University in accordance with its conflict of interest policies.

#### **Contact Information**

Contact Bobbi Woolwine, LCSW at

- if you experience thoughts of suicide or feel you are at risk of harming yourself, or
- if you feel you have had a research-related injury or a bad reaction to the study drug

Contact Dr. Michael Treadway at

- if you have any questions about this study or your part in it, or
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at

- if you have questions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="http://www.surveymonkey.com/s/6ZDMW75">http://www.surveymonkey.com/s/6ZDMW75</a>.

#### Consent

#### TO BE FILLED OUT BY SUBJECT ONLY

| Please print your name, sign, and date below if you agree to be in the study. By signing this consent and authorizatio |
|---|
| form, you will not give up any of your legal rights. We will give you a copy of the signed form to keep. |

| Name of Subject | |
|--------------------------------------------------------|------|
| Signature of Subject (18 or older and able to consent) | <br> |

 IRB Form 04152016 Version Date: 11262019\_Mod20

Emory University IRB IRB use only

Document Approved On: «ApproveDate»


| TO BE FILLED OUT BY STUDY TEAM ONLY |
|---|
| Name of Person Conducting Informed Consent Discussion |
| Signature of Person Conducting Informed Consent Discussion Date |
| TO BE FILLED OUT BY SUBJECT ONLY – CONSENT TO BE CONTACTED VIA TEXT MESSAGE |
| If you are interested, we may send appointment reminders and scheduling information via text message to your mobile phone. All standard data rates would apply. |
| Please indicate below (with your initials) if you are interested in being contacted via text message. |
| I am interested in receiving appointment reminders and scheduling information via text message. |
| I am <b>NOT</b> interested in receiving appointment reminders and scheduling information via text message. |
| TO BE FILLED OUT BY SUBJECT ONLY – CONSENT FOR PARTICIPATION IN MOBILE APPLICATION ASSESSMENTS |
| If you are interested, we may ask you to download a mobile application and complete brief questionnaires and/or behavioral tasks over the course of the study. The mobile app is currently only available for iOS devices. |
| Please indicate below (with your initials) if you are interested in participating in this component of the study. |
| I am interested in completing the mobile app component of this study and have an iOS device. |
| I am <b>NOT</b> interested in completing the mobile app component of this study and/or do not have an iOS device. |
| TO BE FILLED OUT BY SUBJECT ONLY – CONSENT FOR RECONTACT FOR ADDITIONAL SAMPLES |
| If the urine or blood sample we collect is not sufficient for the further testing we may conduct or if we do not ask you to provide a urine or blood sample one of your study visits, we may ask you if you are willing to return to the lab to provide a sample. |
| Please indicate below (with your initials) if you consent to be re-contacted for this purpose. |
| I agree to be re-contacted for an additional blood or urine sample in the future. |
| I do <b>NOT</b> agree to be re-contacted for an additional blood or urine sample in the future. |